CLINICAL TRIAL: NCT04848870
Title: Prevalence and Characteristics of Dental and Periodontal Lesions in Patients With Sjögren's Syndrome. Establishment of a Biological Saliva Collection.
Brief Title: Dental and Periodontal Status of Patients With Sjögren's Syndrome.
Acronym: CB-SJO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210258
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Sjögren Syndrome
Keywords: Sjögren syndrome; tooth wear; gingival recession
MeSH Terms: conditions — Sjogren's Syndrome; Tooth Wear; Gingival Recession

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of salivary samples from Sjögren patients on routine care in the oral medicine department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sjögren patients: Patients in specialized consultations for Sjögren's patients in the oral medicine department of the Charles Foix Hospital AP-HP France
  Interventions: Other: Salivary samples

INTERVENTIONS:
Other: Salivary samples — collection of salivary samples from Sjögren patients on routine care in the oral medicine department.NA

SUMMARY:
Sjögren's syndrome (SS) is a rare chronic systemic autoimmune disease characterized by destruction of the exocrine glands, including the salivary glands.The lack of saliva exposes the patient to dental caries, and dental wear although this has rarely been shown in Sjögren's patients. Moreover, these patients seem to have more inflammation and gingival recession, although this has not been clearly identified in the literature.

Our main objective is to assess the prevalence of dental wear and gingival recession in patients with Sjögren's syndrome by analyzing of the Basic Erosive Wear Examination (BEWE) score for erosions, Basic Erosive Wear Abrasion (BEWA) score for attrition and percentage of sites with periodontal recessions greater than 3 mm in relation to the total number of sites.

Our secondary objectives are to investigate a correlation between the prevalence of dental and gingival wear, gingival inflammation, Decayed, Missing, and Filled Teeth (DMFT) index and (1) salivary parameters and (2) oral quality of life.

The salivary samples will be kept in a biological collection within the URP2496 for later analysis (biological collection CB-SJO).

DETAILED DESCRIPTION:
Sjögren's syndrome (SS) is a rare chronic systemic autoimmune disease characterized by destruction of the exocrine glands, including the salivary glands leading to hyposiala. The lack of saliva exposes the patient to dental caries, and dental wear although this has rarely been described in Sjögren's patients. Moreover, these patients seem to have more inflammation and gingival recession, but not clinical attachment loss, although this has not been clearly identified in the literature.

The present research focuses on the characterization of tooth wear and gingival recession prevalence in patients with Sjögren syndrome. A correlation of this parameters with salivary parameters (Xerostomia Inventory to assess the dryness, unstimulated salivary rate, stimulated salivary rate, pH and buffer capacity) will be assessed.

The salivary samples will be kept in a biological collection within the URP2496 for later cross-sectional research purposes to identify salivary changes associated with increased risk of dental wear, dental caries, periodontal wear or periodontal inflammation (biological collection CB-SJO).

This is a descriptive, prospective, open-label, non-interventional, single-center study with collection of salivary samples (CB-SJO) from a sample of patients with Sjögren's disease as part of the patient's routine care.

Patients will be recruited in the oral medicine department of the AP-HP Charles Foix hospital (Ivry/seine).

The time-line of the research is consistent with the usual patient management in oral medicine department. As Sjogren is a rare disease, we plan an inclusion period of 60 months. There is 60 months (i.e. 5 years) of follow-up, this means a total research duration of 120 months (i.e. 10 years)

ELIGIBILITY:
Inclusion Criteria:

* Patient with Sjögren Syndrome
* Patient > 18 years old
* Patient affiliated to a social security system, beneficiary or beneficiary of a right other than AME
* Patient who speaks and understands French well enough to be able to read and understand the study information note.
* Patient who does not object to his participation in the study

Exclusion Criteria:

- Patient having expressed his opposition to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population consists of patients coming to consult in the oral medicine department of the Hospital of the AP-HP Charles Foix (Ivry/seine), in a specialized consultation for patients with Sjögren Gougerot syndrome created in collaboration with the Reference Center for Rare Immune Auto Diseases (including Sjögren) of the Rheumatology Department of the Bicêtre Hospital.
  And patients followed in the oral medicine department of the AP-HP Charles Foix Hospital (Ivry/Seine) following oral care after the oral assessment at the Sjogren consultation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2032-01-12 (Estimated); Study Completion 2032-01-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dental wear and gingival recession in patients with Sjögren Syndrome | Once a year for 5 years
  BEWE score, BEWA score, Percentage of sites with periodontal recessions greater than 3 mm of the total number of sites

SECONDARY OUTCOMES:
Correlation between the prevalence of dental wear and gingival recession and (1) salivary parameters and (2) oral quality of life | Once a year for 5 years
  OHIP-14 for the oral quality of life assessment; measure of stimulated and unstimulated flow rate, pH and buffer capacity.; measure of the oral dryness through Xerostomia Inventory
Correlation between severity of the gingival inflammation and (1) salivary parameters and (2) oral quality of life. | Once a year for 5 years
  Gingival inflammation assessed using the Bleeding On Probing score
Correlation between severity of carious disease and (1) salivary parameters and (2) oral quality of life | Once a year for 5 years
  Carious disease assessed using the DFMT index

CONTACTS AND LOCATIONS:
Overall Officials: Marjolaine GOSSET, PUPH, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Catherine CHAUSSAIN, PUPH, Study Director — APHP
Locations (1):
- Service de Médecine bucco-dentaire, Ivry-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
The data (age, medical history, medication, dental brushing habits, tobacco consumption, periodontal charting, number of decayed teeth, number of teeth with fillings, number of missing teeth, BEWE score, salivary data, OHIP-14 and Xerostomia Inventory score) will be collected by the investigator on the Orbis medical record or on the paper CRF. They will be transferred by the investigator of the service or a co-investigator of the service on an anonymized excel database and will be sent by secured link for repatriation to the laboratory URP2496.
Supporting Information: Study Protocol